## Metformin in Kidney Disease

NCT02252081

September 26, 2018

## Dysmetabolism of Chronic Kidney Disease and Vascular Health—Aim 2

## **Rationale and Specific Aims for Aim 2**

The ultimate goal of this proposal was to understand the relative and combined impact of obesity and CKD on the generation and maintenance of insulin resistance and their impact on cardiovascular health.

**Specific Aim 2**: To study the effects of metformin, an AMPK activator, on metabolic disturbances associated with obesity and moderate CKD.

- **S.A.2.a:** To test if metformin will improve LAR in obese patients with moderate CKD compared to placebo.
- **S.A.2.b:** To test if metformin will improve markers of systemic inflammation, oxidative stress, endothelial dysfunction (flow mediated vasodilation [FMD] by brachial doppler) in obese patients with moderate CKD compared to placebo.
- **S.A.2.c:** To test if metformin will improve atherosclerosis markers (pulse wave velocity and CIMT) and reduce clinical CVD events in obese patients with moderate CKD compared to placebo.

<u>Hypothesis</u>: We hypothesize that the administration of metformin in obese CKD patients will significantly improve the adipokine profiles—particularly through a reduction in LAR. Additionally, that it will improve systemic inflammation, oxidative stress, and endothelial function (flow mediated vasodilation), which may or may not be mediated by changes in adipokines. Finally, we hypothesize that improvements in these markers of vascular health will translate into reduced arterial stiffness and less clinical CV events.

## **Inclusion/Exclusion Criteria**

There will be no restriction on gender (except pregnant women), race, and age (except less than 18 years old) or disease etiology for patient selection or exclusion except as stated below.

#### Inclusion Criteria:

- 1. Age ≥ 18 years old;
- 2. Ability to give informed consent;
- 3. Life expectancy greater than 6 months;
- 4. Estimated GFR 30-59 ml/min/1.73m<sup>2</sup>;
- 5. Overweight (BMI  $\geq$  25 to < 30 kg/m²) or obese (BMI  $\geq$  30 kg/m²); or normal (BMI  $\geq$  18.5 to < 25 kg/m²) if pre-diabetic or insulin resistant.

## Exclusion Criteria (all subject groups):

- 1. Pregnancy or breast feeding;
- 2. Presence or history of Diabetes Mellitus type I or II
- 3. History of metformin use or any insulin sensitizer or any drug for the treatment of metabolic syndrome over the last one year;
- 4. Any acute kidney injury episode in the last 4 months due to the risk of recurrent AKI;
- 5. Proteinuria of > 5 g in 24 hours determined by a 24 hour urine collection or PCR > 4.5;
- 6. Uncontrolled hypertension with systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 100 mmHg;
- 7. Patients with new changes to their antihypertensive regimen over the last 1 month;
- 8. Severe, unstable, or active inflammatory disease; active infection including seropositive HIV, Hepatitis B or C; active connective tissue disorder; or moderate to severe liver disease;
- 9. Decompensated heart failure:

- 10. Recent hospitalization or surgical procedure within 1 month prior to the study for any cause;
- 11. Current active malignancy or cancer history in the prior 2 years (excluding squamous cell and basal cell skin cancers);
- 12. Known intolerance to the study drug;
- 13. Patient receiving oral or injected steroids;
- 14. Use of any investigational product or device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.

## **Enrollment/Randomization**

All studies will be conducted at the Vanderbilt University Medical Center General Clinical Research Center (GCRC) or at the Nashville VA Tennessee Valley HealthCare System (TVHS). Institutional review board approval have been obtained at both institutions and written informed consent from all study subjects were obtained.

<u>Human Subjects Involvement and Characteristics</u>: We propose to study 120 overweight or obese patients with CKD Stages 3 – 4 for Specific Aim 2. All participants will have a baseline assessment, as well as on-going monitoring, of their health status as documented in their medical record.

## **Study Procedures**

The design is a randomized, double-blind, placebo-controlled study. Once the subject is determined to be eligible, we will randomly assign him/her to metformin versus placebo as depicted in **Figure 11**. The investigators and the study subjects will be blinded to the treatment. Each subject will be treated for 4 months (16 weeks). All of the visits will happen either at the General Clinical Research Center (GCRC) at Vanderbilt University or at the Nashville VA.



Once the baseline studies are completed (see below), we will start the subjects on the randomly assigned protocol of metformin versus matching placebo. The metformin dose will be 1500 mg daily for people with eGFR > 45 ml/min per 1.73 m² and 500 to 1000 mg daily dose for those with an eGFR 30 to  $\leq$  45 ml/min per 1.73 m². All medications and matching placebo will be prepared and dispensed by either Vanderbilt's Investigational Drug Services (IDS) or the VA pharmacy by the investigational drug/pharmacy research team.

**Table. Schedule of Procedures** 

| Procedure | Weeks<br>-2 to 0 | Week<br>0 | Week<br>2 | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>56<br>Optio<br>nal |
|---|---|---|---|---|---|---|---|---|---|
| Vital signs | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Physical exam | ✓ | | | | ✓ | | ✓ | ✓ | ✓ |
| Blood collection | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | | |
| Urine collection | ✓ | ✓ | | ✓ | ✓ | | ✓ | | |
| Urine protein | ✓ | | | | | | | | |
| Urine creatinine | ✓ | | | | | | | | |
| OGTT | | ✓ | | | | | | | |
| CMP (fasting) | ✓ | | | ✓ | ✓ | ✓ | ✓ | | |
| Glycohemoglobin | ✓ | | | | | | | | |
| Lipid panel | ✓ | | | | | | ✓ | | |
| CBC | ✓ | | | | ✓ | | ✓ | | |
| Lactic acid | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | | |
| Serum Pregnancy test | | ✓ | | | | | | | |
| DEXA | | ✓ | | | | | | | |
| Brachial artery Doppler (FMD) | | ✓ | | | | | ✓ | | |
| PWV | | ✓ | | | | | ✓ | | |
| CIMT | | ✓ | | | | | ✓ | | |
| Questionnaires | | ✓ | | | | | ✓ | | |
| LDF (optional) | | ✓ | | | | | ✓ | | |
| Study drug/placebo dispensing | | ✓ | | ✓ | ✓ | ✓ | | | |

**Screening Visit:** Within about two weeks up to the start of the Treatment Phase (which begins at the Baseline Visit) and after the subject has provided informed consent, the subject will be asked to come in fasting state and the following information will be collected:

- Inclusion/exclusion
- Demographics
- Medical history
- Concomitant medications

Also, the following procedures and assessments will be performed:

- Vital signs
- Physical exam (may be performed instead at Baseline Visit)
- If a subject has had a CBC (complete blood count) test within 2 weeks of the stipulated study entry date as part of routine medical care, this value will be counted as the screening value and entry value will be drawn at the Baseline Visit.
- If CBC is drawn for screening, it will be counted as entry value at the Baseline Visit.

- CMP (comprehensive metabolic panel fasting state), liver function test, glycated hemoglobin, and lipid panel
- Urine protein and creatinine

**Baseline Visit (Week 0):** Subjects that qualify for the study will be asked to come in a fasted state. At the Baseline Visit, the following information will be collected:

- Concomitant medications (medication reconciliation)
- Medical history and concurrent illnesses

Also, the following procedures and assessments will be performed:

- Vital signs
- Physical exam (if not obtained at the Screening Visit)
- Lactic acid
- CBC (if not obtained at the Screening Visit) and an optional DNA blood sample
- Serum Pregnancy test
- Dual Energy x-ray absorptiometry (DEXA)
- If CBC is drawn for screening, it will be counted as entry value at the Baseline Visit.
- CMP (comprehensive metabolic panel fasting state), liver function test, glycated hemoglobin, and lipid panel. If drawn for screening, it will be counted as entry value at the Baseline Visit, otherwise they will be drawn at the baseline visit
- Oral glucose tolerance test (OGTT), Brachial artery Doppler (flow mediated dilation of the brachial artery), pulse wave velocity (PWV), and carotid intima-media thickness (CIMT), as well as an optional laser Doppler flowmetry (LDF)
- Blood samples for research labs including study outcomes (inflammatory markers, oxidative stress marker; endothelial function markers; hormones: insulin, leptin, adiponectin/resistin)
- Urine sample for research labs
- Study drug will be dispensed.
- FACIT Fatigue Scale and CESD-10 Questionnaire

**Week 2 Visit:** At the Week 2 Visit, the following information will be collected:

- Concomitant medications
- Adverse Events (AEs)

Also, the following procedures and assessments will be performed:

- Vital signs
- Lactic acid
- Metformin level (not to draw if patient still up-titrating)

Week 4 Visit: At the Week 4 Visit, the following information will be collected:

- Concomitant medications
- Adverse Events (AEs)

Also, the following procedures and assessments will be performed:

- Vital signs
- Lactic acid, CMP and liver function

141513PRO clean 9 26 2018 (short version)

- Study drug will be dispensed.
- Metformin levels

**Week 8 Visit:** At the Week 8 Visit, the following information will be collected:

- Concomitant medications
- Adverse Events (AEs)

Also, the following procedures and assessments will be performed:

- Vital signs
- Physical exam
- Lactic acid, CMP, CBC and liver function
- Blood samples for research labs including study outcomes (inflammatory markers; oxidative stress marker; endothelial function markers; hormones: insulin, leptin, adiponectin/resistin)
- Urine sample for research labs
- Study drug will be dispensed.

Week 12 Visit: At the Week 12 Visit, the following information will be collected:

- Concomitant medications
- Adverse Events (AEs)

Also, the following procedures and assessments will be performed:

- Vital signs
- Lactic acid, CMP and liver function
- Study drug will be dispensed.

Week 16 Visit: At the Week 16 Visit, the following information will be collected:

- Concomitant medications
- Adverse Events (AEs)

Also, the following procedures and assessments will be performed:

- Vital signs
- Physical exam
- Lactic acid, CBC, CMP, lipid panel and liver function
- Brachial artery Doppler (flow mediated dilation), pulse wave velocity (PWV), and carotid intima-media thickness (CIMT), as well as an optional laser Doppler flowmetry (LDF)
- Blood samples for research labs including study outcomes (inflammatory markers; oxidative stress marker; endothelial function markers; hormones: insulin, leptin, adiponectin/resistin)
- Urine sample for research labs
- FACIT Fatigue Scale and CESD-10 Questionnaire

**Early Termination Visit:** Subjects who are withdrawn from the study will be asked to come in for end of study assessments. The information collected at this visit, as well as the procedures and assessments, will be the same as the Week 16 Visit.

**Follow-up Visit 1 (Week 20):** There will be a follow-up visit about 4 weeks after the Treatment Phase. The following information will be collected:

- Concomitant medications
- Adverse Events (AEs)

Also, the following procedures and assessments will be performed:

- Vital signs
- Physical exam

**Follow-up Visit 2 which is optional (Week 56):** There will be a second follow-up visit after about 1 year from starting the Treatment Phase. This could also be completed over a phone call. The following information will be collected:

- Concomitant medications
- Adverse Events (AEs)

Also, the following procedures and assessments will be performed:

- Vital signs
- Physical exam

## Standard Methods (all performed for research purposes only):

**Dual-energy x-ray absorptiometry (DEXA):** We will use DEXA to measure the truncal fat mass percent. During the procedure, subjects will lie on a bed for 10-15 minutes while a scanner X-rays their body fat, lean muscle, and bone masses.

**Oral Glucose Tolerance Test (OGTT):** The oral glucose tolerance test will allow us to estimate the body's ability to metabolize (or break down) glucose. A blood sample will be drawn after an overnight 8-hour fast (to measure initial glucose level), then a 75g glucose solution will be administered orally. Four more blood samples will be collected over the next 2 hours (to measure subsequent glucose levels).

**Brachial Artery Doppler:** The brachial artery Doppler measurement will allow us to evaluate endothelial function (hardening of the medium and large arteries). This will let us know the level of vascular disease (diseases of the blood vessels). This study is not painful and is similar to an ultrasound exam. During the procedure a blood pressure cuff will be placed on the forearm. We will take pictures of the vessel in the arm. We will then pump up the blood pressure cuff. It will remain inflated for 5 minutes. Once released, we will collect more pictures. As an optional procedure, we may then administer a single dose of nitroglycerin (a medicine administered to dilate the vessels) under the tongue. We will take a last set of pictures. Blood pressure will be monitored before giving the nitroglycerin. Taking nitroglycerin is optional. The test can still be performed if nitroglycerin is not taken. This test will take a total of about 45 minutes.

**Aortic Pulse Wave Velocity (PWV):** This test will show us the stiffness of the arteries. This test will be measured with an ultrasound machine by a member of the research team. This test does not involve any shots, radiation or invasive procedures. This will take about 1 hour. Any arrhythmia or a problem with the rate or rhythm of the heartbeat may not allow participation in this test.

**Carotid Intima-media Thickness (CIMT):** This test will allow us to estimate the amount of arteriosclerosis (hardening of the medium and large arteries), which is an indication of the level 141513PRO clean 9 26 2018 (short version)

of vascular disease. This study is not painful and is similar to an ultrasound exam. This test will take about 30 minutes.

Laser Doppler Flowmetry (LDF): This optional test will allow us to estimate blood flow in tissues on a microscopic level. This will let us know the level of vascular disease (diseases of the blood vessels). This study is not painful and is similar to an ultrasound exam. During the procedure a blood pressure cuff will be placed on the forearm. We will take pictures of the vessels in the arm. We will then pump up the blood pressure cuff. It will remain inflated for 4 minutes. Once released, we will collect more pictures. We will also warm a small section of the forearm for 2 minutes. We will collect pictures for about 30 minutes. This test will take a total of about 1 hour.

<u>Safety precautions</u>: In this protocol we have the following safety precautions: 1) We will hold the drug during acute illness. Our temporal stopping criteria are discussed below and will be reinforced at each visit. 2) We will provide patients a 24/7 contact number for questions and concerns. 3) Lactic acid measurements will be obtained with our safety laboratories which will happen at least once a month and as needed.

#### Temporary stopping criteria:

- Patients needing radio-contrast exposure (RCN) for any reason will have their metformin withheld for 48 hours prior to and after the exposure. Drug will be restarted only after a follow up creatinine has been measured and the value considered by the PI to be at baseline.
- Patients will be instructed to stop the medication if for any reason they think they have
  an acute illness of any type, acute respiratory infection, gastrointestinal, nausea,
  vomiting or diarrhea; or if there is the underlying risk of being volume depleted.
  Patients will be asked to contact the study personnel immediately and the PI will decide
  and will be responsible as to when it is safe to re-initiate the drug.

#### Permanent stopping criteria:

A patient will be terminated from the study for any of the following reasons:

- eGFR reaches a value of <30 ml/min per 1.73 m<sup>2</sup> in any of the follow-up laboratory assessments.
- Lactate levels are greater than 3.5 in two measurements.
- There are any adverse events or clinical events that the PI judges increases the risk to the patient.
- If metformin level was above the upper limit even when down titrating.
- There are any signs or symptoms of decline or deterioration of their health status.

# **Statistical Considerations Data Analysis Plan**

Demographic and baseline characteristics will be summarized descriptively by treatment group. Continuous variables will be summarized with mean, median, standard deviation, minimum, and maximum. Categorical variables will be summarized with frequency and percentage. Univariate comparison of the baseline variables will be performed using a Pearson chi-square for categorical variable and non-parametric Mann-Whitney U for continuous variables.

The percent changes in outcome variables from baseline to 16 weeks between the intervention arm and the placebo arm will be compared using either linear mixed effect model (if repeated measures are present for that biomarker) or using an ANCOVA of change if there are only a baseline value and an end off study value. Both outcome variables and baseline values of the outcome variables will be log-transformed—thus exponential of regression coefficient for the interaction term will indicate relative difference in %change from baseline and 16 weeks between groups when using and ANCOVA of change. Using 8-week or 12-week values in analyses is especially helpful when 16-week measures are missing; thus, patients with missing values can be still included in a regression to achieve intent-to-treat principle. There will be two models: 1) 141513PRO clean 9 26 2018 (short version)

unadjusted, 2) fully adjusted which will adjust for unbalanced baseline covariates (not balanced by randomization) and for potential confounders (demographics, baseline eGFR [as a continuous variable], baseline visceral fat [as a continuous variable], etc. The number of covariates in the model will be limited to prevent overfitting the model.

#### **REFERENCES**

- 1. Levey AS, Atkins R, Coresh J, et al. Chronic kidney disease as a global public health problem: approaches and initiatives a position statement from Kidney Disease Improving Global Outcomes. Kidney Int 2007;72:247-59.
- 2. Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med 2004;351:1296-305.
- 3. Hallan SI, Dahl K, Oien CM, et al. Screening strategies for chronic kidney disease in the general population: follow-up of cross sectional health survey. BMJ 2006;333:1047.
- 4. Stenvinkel P, Carrero JJ, Axelsson J, Lindholm B, Heimburger O, Massy Z. Emerging biomarkers for evaluating cardiovascular risk in the chronic kidney disease patient: how do new pieces fit into the uremic puzzle? Clin J Am Soc Nephrol 2008;3:505-21.
- 5. Kershaw E, Flier JS. Adipose tissue as an endocrine organ. J Clin Endocrinol Metab 2004;89:2548-56.
- 6. Hotta K, Funahashi T, Bodkin NL, et al. Circulating concentrations of the adipocyte protein adiponectin are decreased in parallel with reduced insulin sensitivity during the progression to type 2 diabetes in rhesus monkeys. Diabetes 2001;50:1126-33.
- 7. Eikelis N, Lambert G, Wiesner G, et al. Extra-adipocyte leptin release in human obesity and its relation to sympathoadrenal function. American journal of physiology Endocrinology and metabolism 2004;286:E744-52.
- 8. Wallander M, Soderberg S, Norhammar A. Leptin: a predictor of abnormal glucose tolerance and prognosis in patients with myocardial infarction and without previously known Type 2 diabetes. Diabet Med 2008;25:949-55.
- 9. Norata GD, Raselli S, Grigore L, et al. Leptin:adiponectin ratio is an independent predictor of intima media thickness of the common carotid artery. Stroke; a journal of cerebral circulation 2007;38:2844-6.
- 10. Oda N, Imamura S, Fujita T, et al. The ratio of leptin to adiponectin can be used as an index of insulin resistance. Metabolism: clinical and experimental 2008;57:268-73.
- 11. Satoh N, Naruse M, Usui T, et al. Leptin-to-adiponectin ratio as a potential atherogenic index in obese type 2 diabetic patients. Diabetes Care 2004;27:2488-90.
- 12. Chen J, Muntner P, Hamm LL, et al. Insulin resistance and risk of chronic kidney disease in nondiabetic US adults. J Am Soc Nephrol 2003;14:469-77.
- 13. Kobayashi S, Maesato K, Moriya H, Ohtake T, Ikeda T. Insulin resistance in patients with chronic kidney disease. Am J Kidney Dis 2005;45:275-80.
- 14. Pham H, Robinson-Cohen C, Biggs ML, et al. Chronic kidney disease, insulin resistance, and incident diabetes in older adults. Clin J Am Soc Nephrol 2012;7:588-94.
- 15. Nanayakkara PW, Le Poole CY, Fouque D, et al. Plasma adiponectin concentration has an inverse and a non linear association with estimated glomerular filtration rate in patients with K/DOQI 3 5 chronic kidney disease. Clinical nephrology 2009;72:21-30.
- 16. Nordfors L, Lonnqvist F, Heimburger O, Danielsson A, Schalling M, Stenvinkel P. Low leptin gene expression and hyperleptinemia in chronic renal failure. Kidney Int 1998;54:1267-75.
- 17. Aksentijevic D, Bhandari S, Seymour AM. Insulin resistance and altered glucose transporter 4 expression in experimental uremia. Kidney Int 2009;75:711-8.
- 18. Del Prato S, Leonetti F, Simonson DC, Sheehan P, Matsuda M, DeFronzo RA. Effect of sustained physiologic hyperinsulinaemia and hyperglycaemia on insulin secretion and insulin sensitivity in man. Diabetologia 1994;37:1025-35.
- Hung AM, Sundell MB, Egbert P, et al. A comparison of novel and commonly-used indices of insulin sensitivity in African American chronic hemodialysis patients. Clin J Am Soc Nephrol 2011:6:767-74.
- 20. Teta D, Maillard M, Halabi G, Burnier M. The leptin/adiponectin ratio: potential implications for peritoneal dialysis. Kidney Int Suppl 2008:S112-8.
- 21. El Messaoudi S, Rongen GA, de Boer RA, Riksen NP. The cardioprotective effects of metformin. Curr Opin Lipidol 2011;22:445-53.

- 22. Grisouard J, Dembinski K, Mayer D, Keller U, Muller B, Christ-Crain M. Targeting AMP-activated protein kinase in adipocytes to modulate obesity-related adipokine production associated with insulin resistance and breast cancer cell proliferation. Diabetol Metab Syndr 2011;3:16.
- 23. Kendall D, Vail A, Amin R, et al. Metformin in Obese Children and Adolescents: The MOCA Trial. J Clin Endocrinol Metab 2013;98:322-9.
- 24. Knowler WC, Barrett-Connor E, Fowler SE, et al. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med 2002;346:393-403.
- 25. Singh S, Akhtar N, Ahmad J. Plasma adiponectin levels in women with polycystic ovary syndrome: impact of Metformin treatment in a case-control study. Diabetes Metab Syndr 2012;6:207-11.
- 26. Hung AM, Roumie CL, Greevy RA, et al. Comparative effectiveness of incident oral antidiabetic drugs on kidney function. Kidney Int 2012;81:698-706.
- 27. Barsoum RS. Chronic kidney disease in the developing world. N Engl J Med 2006;354:997-9.
- 28. Collins AJ, Foley RN, Chavers B, et al. 'United States Renal Data System 2011 Annual Data Report: Atlas of chronic kidney disease & end-stage renal disease in the United States. Am J Kidney Dis 2012;59:A7, e1-420.
- Longenecker JC, Coresh J, Powe NR, et al. Traditional cardiovascular disease risk factors in dialysis patients compared with the general population: the CHOICE Study. J Am Soc Nephrol 2002;13:1918-27.
- 30. Weiner DE, Tighiouart H, Elsayed EF, et al. The Framingham predictive instrument in chronic kidney disease. J Am Coll Cardiol 2007;50:217-24.
- 31. Smith D, DeFronzo RA. Insulin resistance in uremia mediated by postbinding defects. Kidney Int 1982;22:54-62.
- 32. Rabkin R, Kitaji J. Renal metabolism of peptide hormones. Miner Electrolyte Metab 1983;9:212-26.
- 33. Holmang A, Yoshida N, Jennische E, Waldenstrom A, Bjorntorp P. The effects of hyperinsulinaemia on myocardial mass, blood pressure regulation and central haemodynamics in rats. Eur J Clin Invest 1996;26:973-8.
- 34. Shimizu I, Minamino T, Toko H, et al. Excessive cardiac insulin signaling exacerbates systolic dysfunction induced by pressure overload in rodents. J Clin Invest 2010;120:1506-14.
- 35. Semple D, Smith K, Bhandari S, Seymour A. Uremic Cardiomyopathy and Insulin Resistance: A Critical Role for Akt? . Journal of the American Society of Nephrology 2011;22:207-15.
- 36. DeFronzo RA. Insulin and renal sodium handling: clinical implications. Int J Obes 1981;5 suppl 1:93-104.
- 37. Kadowaki T, Yamauchi T, Kubota N, Hara K, Ueki K, Tobe K. Adiponectin and adiponectin receptors in insulin resistance, diabetes, and the metabolic syndrome. J Clin Invest 2006;116:1784-92.
- 38. Ouchi N, Kihara S, Arita Y, et al. Adiponectin, an adipocyte-derived plasma protein, inhibits endothelial NF-kappaB signaling through a cAMP-dependent pathway. Circulation 2000;102:1296-301.
- 39. Fu Y, Luo N, Klein RL, Garvey WT. Adiponectin promotes adipocyte differentiation, insulin sensitivity, and lipid accumulation. Journal of lipid research 2005;46:1369-79.
- 40. Tao L, Gao E, Jiao X, et al. Adiponectin cardioprotection after myocardial ischemia/reperfusion involves the reduction of oxidative/nitrative stress. Circulation 2007;115:1408-16.
- 41. Kadowaki T, Yamauchi T. Adiponectin and adiponectin receptors. Endocrine reviews 2005:26:439-51.
- 42. Maeda N, Shimomura I, Kishida K, et al. Diet-induced insulin resistance in mice lacking adiponectin/ACRP30. Nature medicine 2002;8:731-7.
- 43. Kubota N, Terauchi Y, Yamauchi T, et al. Disruption of adiponectin causes insulin resistance and neointimal formation. The Journal of biological chemistry 2002;277:25863-6.

- 44. Yamauchi T, Kamon J, Minokoshi Y, et al. Adiponectin stimulates glucose utilization and fatty-acid oxidation by activating AMP-activated protein kinase. Nature medicine 2002:8:1288-95.
- 45. Ouedraogo R, Wu X, Xu SQ, et al. Adiponectin suppression of high-glucose-induced reactive oxygen species in vascular endothelial cells: evidence for involvement of a cAMP signaling pathway. Diabetes 2006;55:1840-6.
- 46. Prior SL, Tang TS, Gill GV, Bain SC, Stephens JW. Adiponectin, total antioxidant status, and urine albumin excretion in the low-risk "Golden Years" type 1 diabetes mellitus cohort. Metabolism: clinical and experimental 2011;60:173-9.
- 47. Lihn AS, Bruun JM, He G, Pedersen SB, Jensen PF, Richelsen B. Lower expression of adiponectin mRNA in visceral adipose tissue in lean and obese subjects. Molecular and cellular endocrinology 2004;219:9-15.
- 48. Takamura N, Hayashida N, Hagane K, et al. Leptin to high-molecular-weight adiponectin ratio is independently correlated with carotid intima-media thickness in men, but not in women. Biomarkers 2010;15:340-4.
- 49. Kiec-Klimczak M, Malczewska-Malec M, Huszno B. [Leptin to adiponectin ratio, as an index of insulin resistance and atherosclerosis development]. Przegl Lek 2008;65:844-9.
- Kappelle PJ, Dullaart RP, van Beek AP, Hillege HL, Wolffenbuttel BH. The plasma leptin/adiponectin ratio predicts first cardiovascular event in men: A prospective nested casecontrol study. Eur J Intern Med 2012.
- 51. Finucane FM, Luan J, Wareham NJ, et al. Correlation of the leptin:adiponectin ratio with measures of insulin resistance in non-diabetic individuals. Diabetologia 2009;52:2345-9.
- 52. Kotani K, Shimohiro H, Sakane N. The relationship between leptin:adiponectin ratio and carotid intima-media thickness in asymptomatic females. Stroke; a journal of cerebral circulation 2008;39:e32-3; author reply e4.
- 53. Inoue M, Yano M, Yamakado M, Maehata E, Suzuki S. Relationship between the adiponectin-leptin ratio and parameters of insulin resistance in subjects without hyperglycemia. Metabolism: clinical and experimental 2006;55:1248-54.
- 54. Park JT, Yoo TH, Kim JK, et al. Leptin/Adiponectin Ratio Is an Independent Predictor of Mortality in Nondiabetic Peritoneal Dialysis Patients. Perit Dial Int 2012.
- 55. Hung AM, Ellis CD, Shintani A, Booker C, Ikizler TA. IL-1beta receptor antagonist reduces inflammation in hemodialysis patients. J Am Soc Nephrol 2011;22:437-42.
- 56. Hung AM, Ikizler TA. Factors determining insulin resistance in chronic hemodialysis patients. Contrib Nephrol 2011;171:127-34.
- 57. Hung A, Pupim L, Yu C, et al. Determinants of C-reactive protein in chronic hemodialysis patients: relevance of dialysis catheter utilization. Hemodialysis international International Symposium on Home Hemodialysis 2008;12:236-43.
- 58. Himmelfarb J, Hakim RM. Oxidative stress in uremia. Current opinion in nephrology and hypertension 2003;12:593-8.
- 59. Ikizler TA, Morrow JD, Roberts LJ, et al. Plasma F2-isoprostane levels are elevated in chronic hemodialysis patients. Clinical nephrology 2002;58:190-7.
- 60. Ramos LF, Shintani A, Ikizler TA, Himmelfarb J. Oxidative stress and inflammation are associated with adiposity in moderate to severe CKD. J Am Soc Nephrol 2008;19:593-9.
- 61. Dounousi E, Papavasiliou E, Makedou A, et al. Oxidative stress is progressively enhanced with advancing stages of CKD. Am J Kidney Dis 2006;48:752-60.
- 62. Himmelfarb J. Linking oxidative stress and inflammation in kidney disease: which is the chicken and which is the egg? Seminars in dialysis 2004;17:449-54.
- 63. Holvoet P, Lee DH, Steffes M, Gross M, Jacobs DR, Jr. Association between circulating oxidized low-density lipoprotein and incidence of the metabolic syndrome. JAMA 2008;299:2287-93.
- 64. Park K, Gross M, Lee DH, et al. Oxidative stress and insulin resistance: the coronary artery risk development in young adults study. Diabetes Care 2009;32:1302-7.

- 65. Annuk M, Zilmer M, Lind L, Linde T, Fellstrom B. Oxidative stress and endothelial function in chronic renal failure. J Am Soc Nephrol 2001;12:2747-52.
- 66. de Aguiar LG, Bahia LR, Villela N, et al. Metformin improves endothelial vascular reactivity in first-degree relatives of type 2 diabetic patients with metabolic syndrome and normal glucose tolerance. Diabetes Care 2006;29:1083-9.
- 67. Kelly T, Yang W, Chen C-S, Reynolds K, He J. Global burden of obesity in 2005 and projections to 2030. Int J Obesity 2008;32:1431-7.
- 68. Lash JP, Go AS, Appel LJ, et al. Chronic Renal Insufficiency Cohort (CRIC) Study: baseline characteristics and associations with kidney function. Clin J Am Soc Nephrol 2009;4:1302-11.
- 69. Fox CS, Massaro JM, Hoffmann U, et al. Abdominal visceral and subcutaneous adipose tissue compartments: association with metabolic risk factors in the Framingham Heart Study. Circulation 2007;116:39-48.
- 70. Kaul S, Rothney MP, Peters DM, et al. Dual-energy X-ray absorptiometry for quantification of visceral fat. Obesity (Silver Spring) 2012;20:1313-8.
- 71. Flegal KM, Kit BK, Orpana H, Graubard BI. Association of all-cause mortality with overweight and obesity using standard body mass index categories: a systematic review and meta-analysis. JAMA 2013;309:71-82.
- 72. Chertow GM, Hsu CY, Johansen KL. The enlarging body of evidence: obesity and chronic kidney disease. J Am Soc Nephrol 2006;17:1501-2.
- 73. Korolczuk A, Dudka J. Increased Risk of Cardiovascular Complications in Chronic Kidney Disease: A Possible Role of Leptin. Curr Pharm Des 2013.
- 74. Hsu CY, McCulloch CE, Iribarren C, Darbinian J, Go AS. Body mass index and risk for end-stage renal disease. Ann Intern Med 2006;144:21-8.
- 75. Wickman C, Kramer H. Obesity and kidney disease: potential mechanisms. Semin Nephrol 2013;33:14-22.
- 76. Wolf G, Ziyadeh FN. Leptin and renal fibrosis. Contrib Nephrol 2006;151:175-83.
- 77. Sharma K. The link between obesity and albuminuria: adiponectin and podocyte dysfunction. Kidney Int 2009;76:145-8.
- 78. Decleves AE, Mathew AV, Cunard R, Sharma K. AMPK mediates the initiation of kidney disease induced by a high-fat diet. J Am Soc Nephrol 2011;22:1846-55.
- 79. Hemmelgarn BR, Manns BJ, Lloyd A, et al. Relation between kidney function, proteinuria, and adverse outcomes. JAMA 2010;303:423-9.
- 80. Viollet B, Guigas B, Sanz Garcia N, Leclerc J, Foretz M, Andreelli F. Cellular and molecular mechanisms of metformin: an overview. Clin Sci (Lond) 2012;122:253-70.
- 81. Klein J, Westphal S, Kraus D, et al. Metformin inhibits leptin secretion via a mitogen-activated protein kinase signalling pathway in brown adipocytes. J Endocrinol 2004;183:299-307.
- 82. Roumie CL, Hung AM, Greevy RA, et al. Comparative effectiveness of sulfonylurea and metformin monotherapy on risk of cardiovascular events in type 2 diabetes mellitus. Ann Intern Med 2012.
- 83. Hung AM, Sundell MB, Plotnikova NE, et al. A Pilot Study of Active Vitamin D Administration and Insulin Resistance in African American Patients Undergoing Chronic Hemodialysis. J Ren Nutr 2012.
- 84. Deger SM, Sundell MB, Siew ED, et al. Insulin Resistance and Protein Metabolism in Chronic Hemodialysis Patients. J Ren Nutr 2012.
- 85. Trirogoff ML, Shintani A, Himmelfarb J, Ikizler TA. Body mass index and fat mass are the primary correlates of insulin resistance in nondiabetic stage 3-4 chronic kidney disease patients. Am J Clin Nutr 2007;86:1642-8.
- 86. Zhou G, Myers R, Li Y, et al. Role of AMP-activated protein kinase in mechanism of metformin action. J Clin Invest 2001;108:1167-74.
- 87. Sanz P. AMP-activated protein kinase: structure and regulation. Current protein & peptide science 2008;9:478-92.
- 88. Sharma K, Ramachandrarao S, Qiu G, et al. Adiponectin regulates albuminuria and podocyte function in mice. J Clin Invest 2008;118:1645-56.

- 89. Yano Y, Hoshide S, Ishikawa J, et al. Differential impacts of adiponectin on low-grade albuminuria between obese and nonobese persons without diabetes. J Clin Hypertens (Greenwich) 2007;9:775-82.
- 90. Lee MJ, Feliers D, Mariappan MM, et al. A role for AMP-activated protein kinase in diabetes-induced renal hypertrophy. American journal of physiology Renal physiology 2007;292:F617-27.
- 91. Hung AM, Roumie CL, Greevy RA, et al. Kidney function decline in metformin versus sulfonylurea initiators: assessment of time-dependent contribution of weight, blood pressure, and glycemic control. Pharmacoepidemiology and drug safety 2013.
- 92. Matsushita K, Mahmoodi BK, Woodward M, et al. Comparison of risk prediction using the CKD-EPI equation and the MDRD study equation for estimated glomerular filtration rate. JAMA 2012;307:1941-51.
- 93. Celik A, Ozcetin M, Celikyay ZR, et al. Evaluation of possible subclinical atherosclerosis in adolescents with a family history of premature atherosclerosis. Atherosclerosis 2012;222:537-40.
- Greenland P, Alpert JS, Beller GA, et al. 2010 ACCF/AHA guideline for assessment of cardiovascular risk in asymptomatic adults: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation 2010;122:e584-636.
- 95. Frid A, Sterner GN, Londahl M, et al. Novel assay of metformin levels in patients with type 2 diabetes and varying levels of renal function: clinical recommendations. Diabetes Care 2010;33:1291-3.
- 96. Salpeter SR, Greyber E, Pasternak GA, Salpeter Posthumous EE. Risk of fatal and nonfatal lactic acidosis with metformin use in type 2 diabetes mellitus. The Cochrane database of systematic reviews 2010:CD002967.
- 97. Voytovich MH, Simonsen C, Jenssen T, Hjelmesaeth J, Asberg A, Hartmann A. Short-term treatment with rosiglitazone improves glucose tolerance, insulin sensitivity and endothelial function in renal transplant recipients. Nephrol Dial Transplant 2005;20:413-8.
- 98. Stewart J, Kohen A, Brouder D, et al. Noninvasive interrogation of microvasculature for signs of endothelial dysfunction in patients with chronic renal failure. Am J Physiol Heart Circ Physiol 2004;287:H2687-96.
- 99. Voytovich MH, Asberg A, Hjelmesaeth J, Jenssen T, Hartmann A. Association between insulin resistance and endothelial dysfunction in renal transplant recipients. Clin Transplant 2006;20:195-9.